CLINICAL TRIAL: NCT03099161
Title: A Phase Ib/II Study to Evaluate the Safety and Tolerability of Preladenant as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced Malignancies
Brief Title: Study of Preladenant (MK-3814) Alone and With Pembrolizumab (MK-3475) in Participants With Advanced Solid Tumors (MK-3814A-062)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The data did not support study endpoints
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3814A-062; MK-3814A-062 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-03-30; First posted 2017-04-04 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-02

CONDITIONS: Neoplasm
Keywords: Advanced Solid Tumor; Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Preladenant 25 mg Twice a Day (BID) (Experimental): During an initial dose evaluation phase, participants received 25 mg of preladenant orally twice a day (BID) on Days 1 through 21 of each 21-day cycle (for a maximum of 35 cycles) until the RP2D could be established. The RP2D was to be established based on the number of dose limiting toxicities (DLTs) at each dose level administered. Participants continued receiving 25 mg of preladenant BID on Days 1 through 21 of each infusion cycle until discontinuation or receiving a maximum of 35 cycles.
  Interventions: Drug: preladenant
- Preladenant 50 mg BID (Experimental): During an initial dose evaluation phase, participants received 50 mg of preladenant orally BID on Days 1 through 21 of each 21-day cycle (for a maximum of 35 cycles) until the RP2D could be established. The RP2D was established based on the number of DLTs at each dose level administered. Participants continued receiving 50 mg of preladenant BID on Days 1 through 21 of each infusion cycle until discontinuation or receiving a maximum of 35 cycles.
  Interventions: Drug: preladenant
- Preladenant + Pembrolizumab (Experimental): During an initial dose evaluation phase, participants received 25 mg of preladenant administered orally BID on Days 1 through 21 in combination with 200 mg pembrolizumab administered as an intravenous (IV) infusion on Day 1 of each 21-day cycle (for a maximum of 35 cycles). Participants continued receiving preladenant 25 mg BID in combination with 200 mg pembrolizumab for each infusion cycle until discontinuation or receiving a maximum of 35 cycles.
  Interventions: Drug: preladenant; Biological: pembrolizumab

INTERVENTIONS:
Drug: preladenant — Administered as an oral capsule BID on Days 1 through 21 of each 21-day cycle
  Other Names: MK-3814A
Biological: pembrolizumab — Administered as IV infusion on Day 1 of each 21-day cycle
  Other Names: KEYTRUDA®; MK-3475
  Arms: Preladenant + Pembrolizumab

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of preladenant (MK-3814A) alone and in combination with pembrolizumab (MK-3475) (pembro) in participants with advanced solid tumors that have not responded to prior therapy. This study will be done in 2 parts. Part 1 will identify and confirm the recommended Phase 2 dose (RP2D) of preladenant when given alone or in combination with pembrolizumab. Part 2 of the study will determine the safety and efficacy of preladenant in combination with pembrolizumab at the RP2D in participants with select solid tumors .

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or pathologically-documented, locally-advanced or metastatic solid tumor for which standard therapy, either does not exist or has been proven ineffective, intolerable or refused by the participant. Each participant must have received at least one and up to five prior lines of cancer treatment regimens, excluding neo-adjuvant, adjuvant, maintenance treatment and surgery
* Has provided a tumor tissue sample (archival or newly obtained core or excisional biopsy of a tumor lesion)
* Has measurable disease per RECIST 1.1
* Has an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Females must not be pregnant
* Female and male participants of reproductive potential must agree to use adequate contraception starting from the first dose of study therapy, throughout the study period, and for up to 120 days after the last dose of study therapy

Exclusion Criteria:

* Has disease that is suitable for local treatment administered with curative intent
* Has received previous treatment with an immunomodulatory agent (e.g, anti- Programmed Cell Death Receptor 1/ Programmed Cell Death Receptor Ligand 1 or anti-cytotoxic T-lymphocyte-associated antigen-4) and was discontinued from treatment due to a Grade 3 or higher immune-related adverse event
* Has received previous treatment with an adenosine A2a receptor antagonist (e.g. CPI-444, HTL1071, PBF-509)
* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks of the first dose of study therapy, or has not recovered to Common Toxicity Criteria for Adverse Events (CTCAE) grade 1 or better from any adverse event
* Is currently participating or has participated in a study with an investigational agent or using an investigational device within 28 days of the first dose of study therapy
* Is currently taking or has taken drugs that interfere with Cytochrome P450 (CYP)3A4 or CYP2C8 or grapefruit and star fruit in diet within 14 days of the first dose of study therapy
* Is currently taking or has taken proton pump inhibitors within 5 days of the first dose of study therapy
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days of the first dose of study therapy
* Is expected to require any other form of systemic or localized antineoplastic therapy while on study
* Has a history of a second malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for 5 years
* Has clinically active central nervous system metastases and/or carcinomatous meningitis
* History of a severe hypersensitivity reaction to treatment with the monoclonal antibody/components of the study drug
* Has an active infection requiring therapy
* History of interstitial lung disease
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* History of active tuberculosis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has received a live-virus vaccine within 30 days of the first dose of study therapy
* Has known Human Immunodeficiency Virus (HIV) (HIV 1 or 2 antibodies) and/or known active and acute Hepatitis B or C infections
* Has known psychiatric or substance abuse disorders that would interfere with the ability to cooperate with the requirements of the study
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
* Has not fully recovered from any effects of major surgery without significant detectable infection
* Has had surgery that required general anesthesia within 2 weeks of the first dose of study therapy
* Has had surgery that required regional/epidural anesthesia within 72 hours of the first dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- START Midwest ( Site 0001), Grand Rapids, Michigan, United States
- Canada (2):
  - Princess Margaret Hospital ( Site 0010), Toronto, Ontario
  - Jewish General Hospital ( Site 0011), Montreal, Quebec
- Israel (2):
  - Rambam Health Care Campus ( Site 0020), Haifa
  - Tel Aviv Sourasky Medical Center ( Site 0021), Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to have 2 parts: a dose escalation/confirmation phase (Part 1) and an expansion phase (Part 2). The expansion phase was not conducted due to early study termination.
Groups:
- Preladenant 25 mg Twice a Day (BID): Participants received 25 mg of preladenant administered by oral capsule BID on Days 1 through 21 of each 21-day cycle. Participants were to receive up to 35 cycles of study treatment.
- Preladenant 50 mg BID: Participants received 50 mg of preladenant administered by oral capsule BID on Days 1 through 21 of each 21-day cycle. Participants were to receive up to 35 cycles of study treatment.
- Preladenant 25 mg BID + Pembrolizumab 200 mg: Participants received 25 mg of preladenant administered by oral capsule BID on Days 1 through 21 and pembrolizumab 200 mg administered by intravenous (IV) infusion on Day 1 of each 21-day cycle. Participants were to receive up to 35 cycles of study treatment.
Period: Overall Study
Arm/Group | Preladenant 25 mg Twice a Day (BID) | Preladenant 50 mg BID | Preladenant 25 mg BID + Pembrolizumab 200 mg
Started | 3 | 4 | 3
Completed | 0 | 0 | 0
Not Completed | 3 | 4 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Progressive Disease | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Preladenant 25 mg BID: Participants received 25 mg of preladenant administered by oral capsule BID on Days 1 through 21 of each 21-day cycle. Participants were to receive up to 35 cycles of study treatment.
- Preladenant 25 mg BID + Pembrolizumab 200 mg: Participants received 25 mg of preladenant administered by oral capsule BID on Days 1 through 21 and pembrolizumab 200 mg administered by IV infusion on Day 1 of each 21-day cycle. Participants were to receive up to 35 cycles of study treatment.
- Total: Total of all reporting groups
Arm/Group | Preladenant 25 mg BID | Preladenant 50 mg BID | Preladenant 25 mg BID + Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 3 | 4 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (10.8) | 40.3 (16.3) | 41.3 (18.5) | 46.9 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 1 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race of participants is presented.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 3 | 4 | 3 | 10
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature; Grade 2: Ambulatory & capable of all self-care but unable to carry out any work activities, up & about >50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair >50% of waking hours; Grade 4: Completely disabled, cannot carry on any self-care, totally confined to bed or chair; or Grade 5: Dead.
  Participants
    ECOG PS=0 | 2 | 2 | 2 | 6
    ECOG PS=1 | 1 | 2 | 1 | 4
Prior Line of Therapy [Count of Participants; unit: Participants] — Participants were required to have an advanced solid tumor that was unresponsive to 1 to 5 lines of prior therapy. The number of prior lines of therapy is presented.
  Participants
    First Line | 2 | 2 | 0 | 4
    Second Line | 0 | 2 | 3 | 5
    Third Line | 0 | 0 | 0 | 0
    Fourth Line | 1 | 0 | 0 | 1
    Fifth Line | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4. A DLT was defined as any of the following events: Grade (Gr) 4 non-hematologic toxicity (not laboratory); Gr 4 hematologic toxicity lasting ≥7 days; Gr 4 thrombocytopenia of any duration; Gr 3 thrombocytopenia with bleeding; Gr 3 non-hematologic toxicity (not laboratory) lasting >3 days despite optimal supportive care; Gr 3 or Gr 4 non-hematologic laboratory value requiring treatment, hospitalization, or persisting for >72 hours; alanine aminotransferase (ALT) or aspartate aminotransferase(AST) >3X upper limit of normal (ULN) WITH total bilirubin >2X ULN with no elevation in alkaline phosphatase (<2X ULN); Febrile neutropenia Gr 3 or 4; discontinuation during Cycle 1 or a >2 week delay in initiating Cycle 2 due to treatment-related toxicity; Missing >25% of preladenant doses as a result of adverse events during Cycle 1; or Gr 5 toxicity.
Time Frame: Cycle 1 (up to 21 days)
Population: All participants who received at least one dose of study treatment in Cycle 1 (21-day Cycle) and were observed for safety or experienced a DLT during Cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Preladenant 25 mg BID | Preladenant 50 mg BID | Preladenant 25 mg BID + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 4 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of the participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 per investigator review. The ORR per RECIST 1.1 for participants is presented.
Time Frame: Up to approximately 8 months
Population: All participants who had a baseline scan that showed measurable disease by investigator assessment and who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Preladenant 25 mg BID | Preladenant 50 mg BID | Preladenant 25 mg BID + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 4 | 3
Percentage of Participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8]

3. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: Up tp approximately 8 months
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Preladenant 25 mg BID | Preladenant 50 mg BID | Preladenant 25 mg BID + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 4 | 3
Participants | 3 | 4 | 3

4. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 8 months
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Preladenant 25 mg BID | Preladenant 50 mg BID | Preladenant 25 mg BID + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 4 | 3
Participants | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to approximately 8 months
Description: The safety population included all participants who received ≥1 dose of study treatment. Per protocol, disease progression of cancer under study was not considered a serious adverse event (SAE) unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded.
Arm/Group | Preladenant 25 mg BID | Preladenant 50 mg BID | Preladenant 25 mg BID + Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/4 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 25 mg BID (N=3) | Preladenant 50 mg BID (N=4) | Preladenant 25 mg BID + Pembrolizumab 200 mg (N=3)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Kidney enlargement (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 25 mg BID (N=3) | Preladenant 50 mg BID (N=4) | Preladenant 25 mg BID + Pembrolizumab 200 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early because the data did not support the study endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT03099161/Prot_SAP_000.pdf